CLINICAL TRIAL: NCT00440050
Title: A Randomized Double-Blind Placebo-Controlled Trial Of The Effects Of Docosahexaenoic Acid (DHA) In Slowing The Progression Of Alzheimer's Disease
Brief Title: DHA (Docosahexaenoic Acid), an Omega 3 Fatty Acid, in Slowing the Progression of Alzheimer's Disease
Acronym: DHA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Collaborators: National Institute on Aging (NIA) (NIH); DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IA0099; 1RC2AG036535 (NIH); ADC-027-DHA
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Results first posted 2010-08-30 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Alzheimer's Disease
Keywords: fish oil; omega-3 fatty acids; EPA
MeSH Terms: conditions — Alzheimer Disease | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. (Experimental): DHA
  Interventions: Drug: DHA (Docosahexaenoic Acid)
- 2. (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DHA (Docosahexaenoic Acid) — 950 mg soft-gel capsules which contain approximately 510 mg DHA, 2 capsules twice a day for 18 months
  Other Names: Neuromins
  Arms: 1.
Drug: Placebo — 2 placebo capsules twice a day for 18 months
  Arms: 2.

SUMMARY:
The purpose of this study is to determine whether chronic DHA (Docosahexaenoic Acid) supplementation slows the progression of cognitive and functional decline in mild to moderate Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Preliminary studies have shown a reduced risk of Alzheimer's disease (AD) in people consuming increased amounts of fish in their diets. Many of the health benefits of fish are attributed to the abundance of omega 3 fatty acids. Docosahexaenoic Acid (DHA) is the most abundant omega 3 fatty acid in the brain. Data from several animal models supports the hypothesis that DHA may be an effective treatment for AD by means of anti-amyloid, antioxidant, and neuroprotectant mechanisms.

In this study, 400 individuals with mild to moderate AD will participate at approximately 53 study sites throughout the US for 18 months. Participants will be randomized so that 60% will receive approximately 2 grams of DHA, divided into 4 capsules, 2 capsules taken twice a day, while 40% receive an identical placebo.

Potential participants will go to their study site for a screening visit, where eligibility is determined, and if accepted, for a baseline visit where cognitive status, behavioral status, functional status, and global severity of dementia will be assessed. Vital signs and biomarker labs will also be obtained. Subsequent visits will occur every three months for medication checks and, every 6 months, further assessments, physical exams, and labs.

Some participants will also take part in MRI (magnetic resonance imaging) and/or CSF (cerebrospinal fluid) sub-studies. For the MRI sub-study, scans will be done prior to beginning the study medication, and again after 18 months. Likewise, for the CSF sub-study, a lumbar puncture will be done prior to beginning the study medication, and again after 18 months.

Enrollment is restricted to individuals who consume no more than 200 mg of DHA per day, which is almost 300% of the average daily intake in an American diet. Individuals who take fish oil or omega 3 fatty acid supplements are also not eligible. Each visit will include completion of a very brief food frequency questionnaire to monitor dietary DHA levels.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 50 years of age or older
* Residing in the community at baseline (includes assisted living facilities, but excludes long-term care nursing facilities)
* MMSE (Mini-Mental State Examination) at screen of 14-26 (inclusive)
* No medical contraindications to study participation
* Fluent in English or Spanish
* Corrected vision and hearing sufficient for compliance with testing procedures
* Supervision available for study medication
* Caregiver/study partner to accompany participant to all visits
* Study partner must have direct contact with the participant more than 2 days/week
* Able to ingest oral medication
* Daily DHA consumption less than or equal to 200 mg/day in prior two months estimated by an abbreviated DHA food frequency questionnaire
* Neuroimaging consistent with the diagnosis of AD at some time after the onset of the memory decline
* Clinical laboratory values must be within normal limits or, if abnormal, must be judged to be clinically insignificant by the investigator
* Stable use of cholinesterase inhibitors and memantine is permitted if doses are stable for 4 months prior to enrollment

Exclusion Criteria:

* Non-AD dementia
* Residence in a long-term care facility at baseline
* History of clinically significant stroke
* Modified Hachinski Ischemia score ≥ 4
* Current evidence or history in past two years of epilepsy, seizure, focal brain lesion, head injury with loss of consciousness or DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition) criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse
* Sensory impairment which would prevent subject from participating in or cooperating with the protocol
* Use of another investigational agent within two months
* Evidence of any significant clinical disorder or laboratory finding that renders the participant unsuitable for receiving an investigational new drug including clinically significant or unstable hematologic, hepatic, cardiovascular (including history of ventricular fibrillation or ventricular tachycardia), pulmonary, gastrointestinal, endocrine, metabolic, renal, or other systemic disease or laboratory abnormality
* Active neoplastic disease (skin tumors other than melanoma may be included; participants with stable prostate cancer may be included at the discretion of the Project Director)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2007-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Quinn, MD, Principal Investigator — Oregon Health and Science University
Locations (51):
- United States (51):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Sun Health Research Institute/Arizona Consortium, Sun City, Arizona
  - University of California Irvine, Irvine, California
  - UCSD Shiley-Marcos Alzheimer's Research Center, La Jolla, California
  - University of Southern California Psychiatry and Behavioral Sciences, Los Angeles, California
  - UCLA Neurology, Los Angeles, California
  - Palo Alto Institute for Research & Education, Palo Alto, California
  - UC-Davis Alzheimer's Disease Center, Sacramento, California
  - Pacific Research Network, San Diego, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center, Dept. of Neurology, Washington D.C., District of Columbia
  - Howard University College of Medicine, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Wien Center, Miami Beach, Florida
  - University of South Florida Suncoast Alzheimer's and Gerontology Center, Tampa, Florida
  - Byrd Alzheimer's Institute, Tampa, Florida
  - Emory University Dept. of Psychiatry, Atlanta, Georgia
  - Northwestern University Cognitive Neurology and Alzheimer Disease Center, Chicago, Illinois
  - Rush Alzheimer's Disease Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Sanders-Brown Center on Aging/Neurology, Lexington, Kentucky
  - Johns Hopkins University Division of Cognitive Neuroscience, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University Alzheimer's Disease Clinical and Research Program, Boston, Massachusetts
  - University of Michigan Dept. of Neurology, Ann Arbor, Michigan
  - Saint Mary's Health Care, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Alzheimer's Disease Research Center, Rochester, Minnesota
  - Saint Louis University, Department of Psychiatry, St Louis, Missouri
  - Washington University ADRC-Memory and Aging Project, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical College, Albany, New York
  - Dent Neurological Institute, Amherst, New York
  - New York University Medical Center, New York, New York
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Mount Sinai School of Medicine, The Bronx, New York
  - Wake Forest University Health Services, Winston-Salem, North Carolina
  - Case Western Reserve University Memory and Aging Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health and Science University Neurology, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Neurology, Providence, Rhode Island
  - Medical University of South Carolina, North Charleston, South Carolina
  - Meharry Medical College, Nashville, Tennessee
  - University of Texas Southwestern-Memory Research Unit, Dallas, Texas
  - Baylor University Department of Neurology, Houston, Texas
  - The Memory Clinic, Bennington, Vermont
  - University of Washington/Seattle Institute for Biomedical & Clinical Research, Seattle, Washington
  - University of Wisconsin Department of Medicine, Madison, Wisconsin

REFERENCES:
- [Background] Horrocks LA, Farooqui AA. Docosahexaenoic acid in the diet: its importance in maintenance and restoration of neural membrane function. Prostaglandins Leukot Essent Fatty Acids. 2004 Apr;70(4):361-72. doi: 10.1016/j.plefa.2003.12.011. PMID 15041028
- [Background] Kalmijn S, van Boxtel MP, Ocke M, Verschuren WM, Kromhout D, Launer LJ. Dietary intake of fatty acids and fish in relation to cognitive performance at middle age. Neurology. 2004 Jan 27;62(2):275-80. doi: 10.1212/01.wnl.0000103860.75218.a5. PMID 14745067
- [Background] Morris MC, Evans DA, Bienias JL, Tangney CC, Bennett DA, Wilson RS, Aggarwal N, Schneider J. Consumption of fish and n-3 fatty acids and risk of incident Alzheimer disease. Arch Neurol. 2003 Jul;60(7):940-6. doi: 10.1001/archneur.60.7.940. PMID 12873849
- [Background] Suzuki H, Morikawa Y, Takahashi H. Effect of DHA oil supplementation on intelligence and visual acuity in the elderly. World Rev Nutr Diet. 2001;88:68-71. doi: 10.1159/000059767. No abstract available. PMID 11935973
- [Background] Calon F, Lim GP, Yang F, Morihara T, Teter B, Ubeda O, Rostaing P, Triller A, Salem N Jr, Ashe KH, Frautschy SA, Cole GM. Docosahexaenoic acid protects from dendritic pathology in an Alzheimer's disease mouse model. Neuron. 2004 Sep 2;43(5):633-45. doi: 10.1016/j.neuron.2004.08.013. PMID 15339646
- [Background] Lim GP, Calon F, Morihara T, Yang F, Teter B, Ubeda O, Salem N Jr, Frautschy SA, Cole GM. A diet enriched with the omega-3 fatty acid docosahexaenoic acid reduces amyloid burden in an aged Alzheimer mouse model. J Neurosci. 2005 Mar 23;25(12):3032-40. doi: 10.1523/JNEUROSCI.4225-04.2005. PMID 15788759
- [Derived] Yassine HN, Rawat V, Mack WJ, Quinn JF, Yurko-Mauro K, Bailey-Hall E, Aisen PS, Chui HC, Schneider LS. The effect of APOE genotype on the delivery of DHA to cerebrospinal fluid in Alzheimer's disease. Alzheimers Res Ther. 2016 Jun 30;8:25. doi: 10.1186/s13195-016-0194-x. PMID 27358067
- [Derived] Quinn JF, Raman R, Thomas RG, Yurko-Mauro K, Nelson EB, Van Dyck C, Galvin JE, Emond J, Jack CR Jr, Weiner M, Shinto L, Aisen PS. Docosahexaenoic acid supplementation and cognitive decline in Alzheimer disease: a randomized trial. JAMA. 2010 Nov 3;304(17):1903-11. doi: 10.1001/jama.2010.1510. PMID 21045096

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 51 sites in the United States between February and November 2007.
Pre-assignment Details: Out of 555 subjects screened, 402 met the study criteria and were randomized.
Groups:
- Placebo: Dosing of 2 grams of placebo administered in a divided dose twice daily with food.
- Docosahexaenoic Acid (DHA): Dosing of 2 grams of DHA administered in a divided dose twice daily with food.
Period: Overall Study
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Started | 164 | 238
Completed | 124 | 171
Not Completed | 40 | 67

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Docosahexaenoic Acid (DHA) | Total
Number analyzed (Participants) | 164 | 238 | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (9.3) | 76 (7.8) | 76 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 112 | 210
  Male | 66 | 126 | 192
Region of Enrollment [Number; unit: participants]
  United States | 164 | 238 | 402

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change on the ADAS-Cog 11.
Description: ADAS-cog 11 = Alzheimer's Disease Assessment Scale, cognitive sub-scale in points per year. This is a psychometric measure sensitive to change in mild to moderate AD. The range of this instrument is 0 to 70 with higher numbers indicating greater impairment.
Time Frame: Baseline, 6, 12, 18 months
Measure: Mean (Standard Deviation); unit: ADAS points per year
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Number analyzed (Participants) | 164 | 238
ADAS points per year | 7.98 (9.84) | 8.27 (8.9)

2. Primary Outcome: Rate of Change on CDR-SOB
Description: CDR-SOB = Clinical Dementia Rating, Sum of Boxes. This is a global rating of dementia severity based on the clinician's interpretation of the history and examination. The range of this instrument is 0 to 18 with higher numbers indicating greater impairment.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Number analyzed (Participants) | 164 | 238
Units on a scale | 2.87 (2.93) | 2.93 (2.83)

3. Secondary Outcome: ADCS-ADL
Description: ADCS-ADL = Alzheimer's Disease Cooperative Study Activities of Daily Living Score. This is a structured questionnaire about activities of daily living, administered to the subject's caregiver/study partner. The range of this instrument is 0 to 6 with lower numbers indicating greater impairment.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Number analyzed (Participants) | 164 | 238
Units on a scale | 10.43 (11.74) | 11.51 (13.23)

4. Secondary Outcome: Neuropsychiatric Inventory (NPI)
Description: The Neuropsychiatric Inventory quantifies behavioral changes in dementia, including depression, anxiety, psychosis, agitation, sleep change, appetite change, and others. This is a structured questionnaire administered to the subject's caregiver/study partner. The range of this instrument is 0 to 120 with higher numbers indicating greater impairment.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Number analyzed (Participants) | 164 | 238
Units on a scale | 2.93 (13.62) | 5.09 (15.08)

ADVERSE EVENTS:
Arm/Group | Placebo | Docosahexaenoic Acid (DHA)
Serious Adverse Events (participants affected / at risk) | 50/164 | 76/238
Other Adverse Events (participants affected / at risk) | 144/164 | 214/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=164) | Docosahexaenoic Acid (DHA) (N=238)
death (General disorders) | 4 (4) | 11/214 (11)
deep venous thrombosis/pulmonary embolus (Blood and lymphatic system disorders) | 2 (2) | 8/214 (8)
other (General disorders) | 44 (44) | 57/214 (57)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=164) | Docosahexaenoic Acid (DHA) (N=238)
diarrhea (Gastrointestinal disorders) | 10 (10) | 18 (18)
urinary tract infection (Renal and urinary disorders) | 12 (12) | 23 (23)
fall (Injury, poisoning and procedural complications) | 33 (33) | 42 (42)
dizziness (General disorders) | 9 (9) | 12 (12)
agitation (Psychiatric disorders) | 12 (12) | 24 (24)
other (General disorders) | 88 (88) | 119 (119)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No